CLINICAL TRIAL: NCT00795288
Title: Effect of Statins on Cerebral Blood Flow After Subarachnoid Hemorrhage
Brief Title: Statins and Cerebral Blood Flow in Subarachnoid Hemorrhage (SAH)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3857 - 54118B
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Subarachnoid Hemorrhage
Keywords: subarachnoid hemorrhage; vasospasm; cerebral blood flow; cerebral metabolism; autoregulation; statin; Vasospasm associated with Subarachnoid hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin, 80 mg/day (Experimental): Simvastatin, 80 mg/day for 21 days
  Interventions: Drug: Simvastatin, 80 mg/day for 21 days
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Simvastatin, 80 mg/day for 21 days — Active treatment group
  Other Names: Simvastatin
  Arms: Simvastatin, 80 mg/day
Drug: placebo — Control group
  Arms: Placebo

SUMMARY:
The primary objective of this project is to investigate the effect of statin therapy on cerebral blood flow in patients with aneurysmal SAH who are randomized to receive or not receive statins in a blinded design.

DETAILED DESCRIPTION:
We will determine if statin therapy improves CBF in patients with aneurysmal subarachnoid hemorrhage. This improvement, if present, may be due to improved basal CBF, improved autoregulatory function, or a mitigation of large arterial narrowing. The information gain from this study will help us to better understand the mechanism of action of statins. This knowledge may be useful in the design of future studies with statins and in the development of other therapies aimed at similar mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* SAH from ruptured cerebral aneurysm within 48 hours of admission.
* Modified Fisher grade 2,3,or 4
* Planned surgical or endovascular aneurysm repair

Exclusion Criteria:

* Pregnancy
* SAH secondary to traumatic or mycotic aneurysms
* Pre-ictal statin therapy
* Contraindication to stain therapy
* WFNS grade 5
* Contraindications to MAP elevation on day 7-10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2008-08; Primary Completion 2013-02 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Diringer, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington Univeristy, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Diringer MN, Dhar R, Scalfani M, Zazulia AR, Chicoine M, Powers WJ, Derdeyn CP. Effect of High-Dose Simvastatin on Cerebral Blood Flow and Static Autoregulation in Subarachnoid Hemorrhage. Neurocrit Care. 2016 Aug;25(1):56-63. doi: 10.1007/s12028-015-0233-7. PMID 26721259

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo; Simvastatin: All SAH patients admitted to our institution were screened for enrollment. The inclusion criteria are as follows: age > 18, SAH from a ruptured cerebral aneurysm enrolled within 48 hours of hemorrhage, modified Fisher grade 2, 3, or 4 on initial CT scan and planned surgical or endovascular aneurysm repair. Patients were randomized to receive either 80 mg of simvastatin or placebo once a day for 21 days after their hemorrhage.
Period: Overall Study
Arm/Group | Placebo | Simvastatin
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Simvastatin: Simvastatin, 80 mg/day
  Simvastatin, 80 mg/day for 21 days: Active treatment group
- Control: placebo: Control group
- Total: Total of all reporting groups
Arm/Group | Simvastatin | Control | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 21 | 42
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (12) | 60 (10) | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 9 | 7 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 19 | 18 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Resting Cerebral Blood Flow During Peak Period of Vasospasm Risk
Description: Resting cerebral blood flow during peak period of vasospasm risk measured by PET
Time Frame: 7-10 days after hemorrhage
Population: Of the total population enrolled complete data sets were available on 25. This was due to patient refusal to perform the PET study, logistical difficulties and technical problems.
  be completed in seven due to logistical difficulties (n = 4) or patient refusal (n = 3). Two of the completed studies could not be analyzed for technical reasons
Measure: Mean (Standard Deviation); unit: mL/100 g/min
Groups:
- Simvastatin: Simvastatin, 80 mg/day once daily for a total of 21 days following acute SAH: Active treatment group Patients were randomized to receive either 80 mg of simvastatin or placebo once a day for 21 days after their hemorrhage.
- Control: placebo: Control group Patients were randomized to receive either 80 mg of simvastatin or placebo once a day for 21 days after their hemorrhage.
Arm/Group | Simvastatin | Control
Number analyzed (Participants) | 13 | 12
mL/100 g/min | .34 (0.1) | .30 (.18)

2. Primary Outcome: Cerebral Autoregulation During Peak Period of Vasospasm Risk
Description: Fraction of patients with impaired static autoregulation (% change in MAP/% change in CVR) * 100 A value of <60 is considered abnormal.
Time Frame: 7-10 days after hemorrhage
Measure: Number; unit: participants
Arm/Group | Simvastatin | Control
Number analyzed (Participants) | 13 | 12
participants | 2 | 2

3. Secondary Outcome: Impact of Statin on Oxygen Extraction Fraction and Cerebral Metabolism During Peak Period of Vasospasm Risk
Description: Oxygen extraction fraction (OEF) is the ratio of Oxygen delivery (ml/100 g/min) and oxygen utilization (ml/100 g/min). It describes the fraction of the oxygen that reaches the brain that it actually uses for energy production.
Time Frame: 7-10 days after hemorrhage
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Simvastatin, 80 mg/Day | Placebo
Number analyzed (Participants) | 13 | 12
ratio | .34 (.1) | .3 (.18)

ADVERSE EVENTS:
Arm/Group | Simvastatin | Control
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No